CLINICAL TRIAL: NCT03844178
Title: Role of Pupil Centroid Shift Compensation on Lower and Higher Order Aberrations During Photorefractive Keratectomy: An Eye-to-Eye Study
Brief Title: Pupil Centroid Shift Compensation in Photorefractive Keratectomy Candidates
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of ophthalmic research center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 97362
Record Dates: First submitted 2019-02-02; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Pupil Centroid Shift
MeSH Terms: interventions — Photorefractive Keratectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The right eyes with compensation for Pupil centroid shift (Active Comparator)
  Interventions: Procedure: The option for compensation of Pupil centroid shift was ON; Drug: installation of Tetracaine 1%; Procedure: Photorefractive keratectomy (PRK)
- The left eyes without compensation for Pupil centroid shift (Active Comparator)
  Interventions: Procedure: The option for compensation of Pupil centroid shift was OFF; Drug: installation of Tetracaine 1%; Procedure: Photorefractive keratectomy (PRK)

INTERVENTIONS:
Procedure: The option for compensation of Pupil centroid shift was ON — The option for compensation of Pupil centroid shift was ON
  Arms: The right eyes with compensation for Pupil centroid shift
Procedure: The option for compensation of Pupil centroid shift was OFF — The option for compensation of Pupil centroid shift was OFF
  Arms: The left eyes without compensation for Pupil centroid shift
Drug: installation of Tetracaine 1% — installation of Tetracaine 1%
Procedure: Photorefractive keratectomy (PRK) — periorbital skin will be prepared with povidone iodine 5%. Iris registration will be performed in all eyes before epithelial removal. Ethylalcohol 20.0% into a 9.0 mm well for 20 seconds will be applied on the central cornea, and then the epithelium of the central 9.0 mm area will be removed by hockey knife. Excimer laser ablation will be performed by Wavelight Allegretto EX500 (Alcon, Fort Worth, TX, USA)

SUMMARY:
patients who are candidates of PRK will be recruited in this intrasubject randomized clinical trial. Inclusion criteria are myopia or myopic astigmatism with refractive cylinder. Exclusion criteria were unstable refractive error, age less than 21 years old, corneal opacity, keratoconus, keratoconus suspects, residual corneal stromal thickness less than 350 µm, moderate or severe dry eye disease and any other ocular pathology other than refractive error. Complete eye exam will be performed preoperatively including: uncorrected distance visual acuity (UDVA), best spectacle corrected distance visual acuity (CDVA), cyclorefraction, slit lamp biomicroscopy, Goldmann applannation tonometry, dual scheimpflug tomography (Ziemmer), topography in mesopic condition accompanied by pupilometry and iris registration (Topolyzer Vario, Alcon Laboratories, Inc., Fort Worth, TX), and funduscopy with dilated pupil.

Surgical Technique The same surgeon (A.F.) will perform all surgeries. After installation of Tetracaine 1%, periorbital skin will be prepared with povidone iodine 5%. Iris registration will be performed in all eyes before epithelial removal. Ethylalcohol 20.0% into a 9.0 mm well for 20 seconds will be applied on the central cornea, and then the epithelium of the central 9.0 mm area will be removed by hockey knife. In the right eye of each patient PCS compensation will be turned on (PCS-On group) and in the left eye it will be turned off (PCS-Off group). Excimer laser ablation will be performed by Wavelight Allegretto EX500 (Alcon, Fort Worth, TX, USA). Selection of which eye to be first ablated will be done randomly. Randomization will be performed based on a computer software by a Biostatistician which produced the first eye to be operated. Static cyclotorsion compensation will be active in all eyes. The ablation profile will be wavefront-optimized in all cases.

Postoperative Course Postoperatively, chloramphenicol 0.5% eye drops and betamethasone 0.1% eye drops will be prescribed every 6 hours for 10 days. Thereafter, Fluorometholone 0.1% eye drops every 6 hours for 1 month and every 8 hours for the next month will be given. Follow-up examinations were scheduled at 1, 2, 3, 4, 7 and 15 days and 1, 2, 3, and 6 months postoperatively. After contact lens removal each follow-up examination includes the UDVA, manifest refraction, and IOP measurements as well as a slit lamp biomicroscopy. Corneal imaging with Galilei tomography, CDVA and cyclorefraction will be performed at the final follow-up examination 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* myopia
* myopic astigmatism

Exclusion Criteria:

* unstable refractive error, age less than 21 years old
* corneal opacity
* keratoconus, keratoconus suspects
* residual corneal stromal thickness less than 350 µm
* moderate or severe dry eye disease
* any other ocular pathology other than refractive error

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-02-10 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative refractive error | 2 months
  Snellen chart and subjective refraction

SECONDARY OUTCOMES:
Root Mean Square (RMS) of higher order aberration | 6 months
  wavefront analysis by galilei scan

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Iran